CLINICAL TRIAL: NCT00026468
Title: Chemoprevention of Duodenal Polyps in Familial Adenomatous Polyposis
Brief Title: Exisulind in Preventing Polyps in Patients With Familial Adenomatous Polyposis
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Principle Investigator has left the University.
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: CDR0000069032; R01CA080852 (NIH); P30CA042014 (NIH); UUMC-IRB-5999-96; NCI-H01-0079
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Colorectal Cancer; Small Intestine Cancer
Keywords: colon cancer; rectal cancer; small intestine cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — sulindac sulfone

INTERVENTIONS:
Drug: exisulind

SUMMARY:
RATIONALE: Exisulind may be effective in preventing the development and growth of polyps in patients who have familial adenomatous polyposis.

PURPOSE: Randomized phase II/III trial to determine the effectiveness of exisulind in preventing the development and growth of polyps in patients who have familial adenomatous polyposis.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the ability of exisulind to inhibit growth and development of duodenal adenomas in patients with familial adenomatous polyposis.
* Determine the effect on apoptosis in polyp vs mucosal tissue in these patients when treated with this drug.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive oral exisulind 4 times daily.
* Arm II: Patients receive oral placebo 4 times daily. Treatment continues for 1 year.

PROJECTED ACCRUAL: A total of 100 patients (50 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following diagnosis:

  * Diagnosis of familial adenomatous polyposis

    * Prior total or subtotal colectomy
  * Attenuated adenomatous polyposis coli

    * May have colon intact
* 10-40 duodenal polyps from second portion to 10 cm distal to papilla of Vater

PATIENT CHARACTERISTICS:

Age:

* 18 to 80

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Hemoglobin at least 10 g/dL
* Platelet count at least 100,000/mm^3
* No active hematologic disease

Hepatic:

* AST and ALT less than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase less than 1.5 times ULN
* No active hepatic disease

Renal:

* Creatinine less than 1.5 mg/dL
* No active renal disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active peptic ulcer disease
* No serious underlying medical or psychiatric illness that would preclude completion of the study or limit survival
* No prisoners or institutionalized patients
* No known allergy to sulindac or related compounds
* No active internal malignancy within the past 5 years
* No alcohol or drug abuse within the past 5 years

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Other:

* No prior non-steroidal anti-inflammatory drugs (NSAIDs) or salicylates more than 10 days a month for the past 3 months
* No concurrent NSAIDs (e.g., mesalamine, olsalazine, azodisalicylate, salsalate, sulfasalazine)
* Aspirin for cardiac reasons allowed (81 mg/day or 325 mg twice/week)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1999-07; Primary Completion 1999-07 (Actual); Study Completion 1999-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A. DiSario, MD, Study Chair — University of Utah